CLINICAL TRIAL: NCT00803933
Title: Phase II b Trial of DB289 for the Treatment of Stage I African Trypanosomiasis
Brief Title: Trial of DB289 for the Treatment of Stage I African Trypanosomiasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immtech Pharmaceuticals, Inc (Industry)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Christian Burri, Study Director, Swiss Tropical Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 289-C-006
Record Dates: First submitted 2008-12-04; First posted 2008-12-08 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-12

CONDITIONS: African Trypanosomiasis
Keywords: first stage; Trypanosoma brucei gambiense; T. b. gambiense; sleeping sickness; First stage T. b. gambiense sleeping sickness
MeSH Terms: conditions — Trypanosomiasis, African | interventions — Pentamidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DB289 (Experimental): Pafuramidine maleate (DB289), 100 mg BID orally
  Interventions: Drug: DB289
- Pentamidine (Active Comparator): Pentamidine isethionate (Aventis) for injection (200 mg/vial), 4 mg/kg QD IM
  Interventions: Drug: Pentamidine

INTERVENTIONS:
Drug: DB289 — Pafuramidine maleate (DB289), 100 mg BID orally
  Other Names: pafuramidine maleate
  Arms: DB289
Drug: Pentamidine — Pentamidine isethionate (Aventis) for injection (200 mg/vial), 4 mg/kg QD IM
  Arms: Pentamidine

SUMMARY:
Human African Trypanosomiasis or sleeping sickness has made a spectacular return during the last decade, and in many places the demand largely surpasses the capacities of the treatment centers. Treatment of the disease remains unsatisfactory. All currently used drugs must be administered parenterally, treatment is lengthy, and adverse drug reactions frequent. There are currently no drugs that are easily administered and have low toxicity, and might thus be used as tools to support disease control.

This study aims to compare the safety and efficacy of DB289, a new, orally administered dication prodrug to pentamidine i.m. injection for the treatment of first stage sleeping sickness. The project will be executed in the framework of an international consortium consisting of several partners from academia, industry and from the Democratic Republic of Congo Ministries of Health.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has early stage T. b. gambiense infection i.e. parasitologically confirmed infection in the blood or lymph node aspirate and greater than or equal to 5 WBC mm-3 detected in the CSF by microscopic examination
2. Patient is 15 to 50 years old
3. Patient has a minimal weight of 35 kilograms
4. If the patient is female of child bearing potential (a women will be considered of non-child bearing potential only if she has been post menopausal for over 2 years or has had a hysterectomy):

   1. she is not lactating,
   2. she had a negative urine pregnancy test result within 24 hours prior to DB289 treatment and
   3. she agrees to use a medically proven method of contraception (abstinence from sexual intercourse is an acceptable method) from the day of consent on until the end of the observation period (day 7).
5. Patient has understood and signed the Informed Consent. If the patient is minor, a legal guardian has signed the Informed Consent

Exclusion Criteria:

1. The patient has late stage T.b. gambiense infection i.e. presence of parasite in the CSF upon microscopic examination or a WBC count of > 5mm-1
2. Active clinically relevant medical conditions that in the Investigator opinion may jeopardize subject safety or interfere with participation in the study, including but not limited to: significant liver diseases, chronic pulmonary diseases, significant cardiovascular diseases, diabetes, thyroid diseases, gout, infection including known HIV infection, CNS trauma or seizure disorders (A list of typical signs and symptoms is provided for guidance of the investigator in attachment 1)
3. Coma Score of less than 9 on the Glasgow Coma Scale (Appendix 8)
4. Withdrawal of consent at any time during the study
5. Any condition which compromises ability to communicate with the investigator as required for the completion of this study.
6. The subject has been previously treated for African Trypanosomiasis.
7. The subject has been previously enrolled in the study. -

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 111 (Actual)
Dates: Start 2003-02; Primary Completion 2004-02 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint was the parasitological cure at 3 months after completion of treatment. | 3 months
The primary outcome measure for safety analysis was the rate of occurrence of Grade 3 or higher adverse events during the observation period. | 12 day

SECONDARY OUTCOMES:
The secondary outcome measure was the incidence rate of adverse events (all Grades combined) during the 7- to 9-day observation period in Treatment Sequence 1 and during the 12-day observation period in Treatment Sequence 2. | 12 day
The number and percentage of subjects with parasitological cure, subjects with confirmed (parasitological) treatment failure, and subjects with suspected treatment failure at 6, 12, and 24 months after completion of treatment. | 6, 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Victor Kande, MD, Principal Investigator — Programme Nationale de Lutte contre la Trypanosomiase Humaine Africaine
Locations (2):
- Republic of the Congo (2):
  - CDTC Maluku, Gombé, Kinshasa
  - Vanga Hospital, Gombé, Kinshasa

REFERENCES:
- [Derived] Burri C, Yeramian PD, Allen JL, Merolle A, Serge KK, Mpanya A, Lutumba P, Mesu VK, Bilenge CM, Lubaki JP, Mpoto AM, Thompson M, Munungu BF, Manuel F, Josenando T, Bernhard SC, Olson CA, Blum J, Tidwell RR, Pohlig G. Efficacy, Safety, and Dose of Pafuramidine, a New Oral Drug for Treatment of First Stage Sleeping Sickness, in a Phase 2a Clinical Study and Phase 2b Randomized Clinical Studies. PLoS Negl Trop Dis. 2016 Feb 16;10(2):e0004362. doi: 10.1371/journal.pntd.0004362. eCollection 2016 Feb. PMID 26881924